CLINICAL TRIAL: NCT04423237
Title: Identification of Risk Factors and Measures to Prevent Liver and Pancreas Complications in Pediatric Patients Undergoing a Hematopoietic Stem Cell Transplant (HSCT)
Brief Title: Risk Factors and Measures to Prevent Liver and Pancreas Complications in Pediatric Patients After HSCT
Status: Completed | Type: Observational
Sponsor: University of Pisa (Other)
Collaborators: IRCCS Burlo Garofolo (Other); University of Genova (Other)
Responsible Party: Principal Investigator, Antonello Di Paolo, M.D., Ph.D., Associated Professor, University of Pisa
Other Study IDs: 1105/2015
Record Dates: First submitted 2020-05-30; First posted 2020-06-09 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Iron Overload
Keywords: iron overload; deferasirox; children; HSCT; toxicity; ductopenia
MeSH Terms: conditions — Iron Overload | interventions — Deferasirox

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Severe Iron Overload (SIO): Children affected by Severe Iron Overload who received DEFERASIROX
  Interventions: Drug: Deferasirox
- Severe Iron Overload + Ductopenia (SIO+D): Children affected by Severe Iron Overload + Ductopenia who received DEFERASIROX
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox — DEFERASIROX administered as per clinical practice and according to technical note
  Other Names: Exjade or Deferasirox Milan

SUMMARY:
Hematopoietic Stem Cell Transplantation (HSCT) is currently a standard procedure for a wide range of blood-oncological diseases and genetic disorders. Recent improvements in transplant technologies, infection prevention and graft-versus-host-disease (GVHD) management procedures have significantly reduced the transplant-related mortality (TRM). However, approximately 50% of pediatric patients may develop liver dysfunction before HSCT and 74% to 85.5% after HSCT, with a TRM related to liver dysfunction reaching 46%. The liver and pancreas complications still remain too high for the difficulties and diagnostic inefficiencies and, consequently, for the lack of targeted and safer therapies. The diagnostic problems can be summarized in 3 major points: a) the histological examination of liver and pancreas parenchyma cannot be routinely performed because of the organ anatomy and the relative risk of the bioptic procedures; b) the lack of specific biomarkers or advanced imaging techniques appropriate for the diagnosis of HSCT complications; c) the multifactorial causes of organ complications, as well as drug toxicities, GVHD, siderosis, ductopenia (considered as an index of hepatic GVHD), the accumulation of potentially toxic substances favored by siderosis and ductopenia. In more than 50% of HSCT patients, siderosis and/or ductopenia may represent common pathological conditions. Furthermore, international guidelines issued by onco-hematology and transplantation scientific societies recommend a chelating treatment with deferasirox in all hematological and oncological patients undergoing an intense transfusion regimen. However, in the presence of siderosis and marked ductopenia, patients receiving deferasirox may experience both severe renal and hematological toxicities and lack of effectiveness of the chelating treatment.

Therefore, the principal aim of the present retrospective study will be the evaluation of the transplant-related mortality (TRM) in patients requiring a chelation treatment according to the Italian guidelines in pediatric patients

DETAILED DESCRIPTION:
The present retrospective study will be conducted at the Bone Marrow Transplant Center, IRCCS Burlo Garofolo, Trieste, Italy. All pediatric patients who underwent one or more allogeneic HSCTs between 2010 and 2018 will be enrolled according to inclusion/exclusion criteria.

The following data will be collected in a retrospective manner:

* Data on the underlying disease (diagnosis, therapeutic protocol, transfusion regimen, possible relapses, type of transplant, conditioning regimen, infectious complications, immunosuppressive treatment, including use of steroids);
* Pre-transplant liver and pancreatic function, as well as quantification of iron content by nuclear magnetic resonance (MRI);
* Pre-transplant histological evaluation of liver parenchyma in case of pre-existing liver disease;
* Post-transplant liver and pancreatic function and the evaluation of parenchymal accumulation of Fe+;
* Length and doses of DFX treatment, and corresponding drug plasma concentrations as per routine drug monitoring protocols;
* Treatment tolerability according to CTC-AE grading V5.0, November 27, 2017 The post-transplant data will be collected within 2 years from HSCT (or the last HSCT when more than one).

The data entered in an appropriate anonymous database will be processed by descriptive statistics and uni- multivariate statistical analyses according to study endpoints. DFX plasma concentrations will be analyzed by means of to a nonlinear mixed effect modeling approach to elaborate a population pharmacokinetic (POP/PK) model. POP/PK findings will be further analyzed together with clinical and laboratory data.

ELIGIBILITY:
Inclusion Criteria:

* one or more allogeneic HSCT
* any type of disease (blood-oncological or genetic), from any type of donor (sibling, MUD, haploidentical) and with any source of stem cells (spinal cord, peripheral blood stem cells, cord blood)
* diagnosis of moderate-to-severe siderosis (by nuclear magnetic resonance imaging, MRI) and who needed a chelation treatment with deferasirox
* one or more liver biopsies in the post-transplant period to perform histological examinations
* Complete results from lab analyses
* 2-year follow-up after HSCT
* therapeutic drug monitoring (TDM) protocol for deferasirox plasma concentration as per clinical routine
* Sign of the informed consent by the parents or legal representatives

Exclusion Criteria:

* Lack of liver biopsies after transplantation, results from laboratory analyses or TDM or MRI
* Lack of informed consent

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric inpatients who a) underwent a HSCT at the Bone Marrow Transplant Center, IRCCS Burlo Garofalo, and b) had a ≥2-year follow-up after transplant. All procedures were performed according to clinical routine protocols
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Transplant-related mortality (TRM) | 0-24 months after transplant
  TRM in SIO/SIO+D patients treated with deferasirox as per Italian guidelines

SECONDARY OUTCOMES:
Post-HSCT liver and pancreatic complications | 0-24 months after transplant
  Incidence of post-HSCT liver and pancreatic complications in SIO/SIO+D patients treated with deferasirox as per Italian guidelines
Time to iron concentration normalization | 0-24 months after transplant
  The times required for the normalization of the Iron Concentration in SIO and SIO+D patients
Statistical analysis of risk factors for ductopenia | 0-24 months after transplant
  The correlation between ductopenia and potential risk factors will be investigated by uni- and multi-variate analyses. The following data will be included in the analyses as potential risk factors: chemo-radiotherapy regimens prior to HSCT (drugs and doses), number of blood transfusions
Minimum plasma concentrations of deferasirox | 0-24 months after transplant
  In SIO/SIO+D patients, a factorial analysis for mixed data and a nonlinear mixed effect modeling approach will be used to investigate plasma pharmacokinetics of deferasirox in terms of patients' exposure (minimum plasma concentration, Cmin) and to evaluate the effect of identified covariates on drug disposition.
Correlation of minimum plasma concentrations of deferasirox with drug tolerability | 0-24 months after transplant
  In SIO/SIO+D patients, uni- and multi-variate analyses will be adopted to assess the correlation of Cmin with treatment tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Maximova, MD, Study Director — Institute for Maternal and Child Health, IRCCS Burlo Garofalo, Trieste, Italy
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Italy

REFERENCES:
- [Background] Maximova N, Zanon D, Pascolo L, Zennaro F, Gregori M, Grosso D, Sonzogni A. Metal accumulation in the renal cortex of a pediatric patient with sickle cell disease: a case report and review of the literature. J Pediatr Hematol Oncol. 2015 May;37(4):311-4. doi: 10.1097/MPH.0000000000000322. PMID 25811747
- [Result] Galeotti L, Ceccherini F, Fucile C, Marini V, Di Paolo A, Maximova N, Mattioli F. Evaluation of Pharmacokinetics and Pharmacodynamics of Deferasirox in Pediatric Patients. Pharmaceutics. 2021 Aug 11;13(8):1238. doi: 10.3390/pharmaceutics13081238. PMID 34452199